CLINICAL TRIAL: NCT04172727
Title: Subarachnoid Block With Ultrasound-Guided Transversalis Fascia Plane Block for Cesarean Sections: A Randomized Placebo-Controlled Double-Blind Study
Brief Title: Subarachnoid Block With Ultrasound-Guided Transversalis Fascia Plane Block for Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AUTF ANESTHESIAOBSTETRIC
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Caesarean Section; Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided transversalis fascia plane block (Active Comparator): 20 mL of 0.25% bupivacaine
  Interventions: Drug: Bupivacaine Hcl 0.25% Inj
- ultrasound guided sham block (Placebo Comparator): 20 mL of saline
  Interventions: Drug: saline 0.9%

INTERVENTIONS:
Drug: Bupivacaine Hcl 0.25% Inj — ultrasound-guided bilateral TFP block with 20 mL of 0.25% bupivacaine
  Arms: ultrasound guided transversalis fascia plane block
Drug: saline 0.9% — ultrasound-guided bilateral TFP block with 20 mL of saline 0.9%
  Arms: ultrasound guided sham block

SUMMARY:
Postoperative pain management is critical for the fulfillment of the maternal duties. The transversalis fascia plane (TFP) block provides adequate postoperative analgesia in the T12 and L1 dermatomes. The aim of this study was to investigate the effect of the TFP block on postoperative opioid consumption and pain scores in patients undergoing cesarean section (CS) under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 45
* American Society of Anesthesiologists (ASA) physical score I or II

Exclusion Criteria:

* Patients who received general anesthesia
* hypersensitivity to the agents to be used
* body mass index (BMI) greater than 35 kg/m2
* coagulopathy
* local infections
* opioid addiction
* pregnancy-related hypertension or diabetes mellitus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women aged between 18 and 45 with American Society of Anesthesiologists (ASA) physical score I or II undergoing elective CS
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
opioid consumption | Postoperative first 24hour
  morphine consumption first 24hour

SECONDARY OUTCOMES:
pain scores | postoperative 0-24 hours
  Visual Analogue Scale (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Ali Ahıskalıoğlu, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serifsoy TE, Tulgar S, Selvi O, Senturk O, Ilter E, Peker BH, Ozer Z. Evaluation of ultrasound-guided transversalis fascia plane block for postoperative analgesia in cesarean section: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2020 Feb;59:56-60. doi: 10.1016/j.jclinane.2019.06.025. Epub 2019 Jun 27. PMID 31255890
- [Background] Hebbard PD. Transversalis fascia plane block, a novel ultrasound-guided abdominal wall nerve block. Can J Anaesth. 2009 Aug;56(8):618-20. doi: 10.1007/s12630-009-9110-1. Epub 2009 Jun 4. No abstract available. PMID 19495909
- [Derived] Aydin ME, Bedir Z, Yayik AM, Celik EC, Ates I, Ahiskalioglu EO, Ahiskalioglu A. Subarachnoid block and ultrasound-guided transversalis fascia plane block for caesarean section: A randomised, double-blind, placebo-controlled trial. Eur J Anaesthesiol. 2020 Sep;37(9):765-772. doi: 10.1097/EJA.0000000000001222. PMID 32412986